CLINICAL TRIAL: NCT04410133
Title: An Open-label, Single-arm, Single-dose, Prospective, Multicenter Phase 3 Study to Establish the Diagnostic Performance of 18F-Fluciclovine Positron Emission Tomography (PET) in Detecting Recurrent Brain Metastases After Radiation Therapy
Brief Title: Study to Establish the Diagnostic Performance of 18F Fluciclovine PET in Detecting Recurrent Brain Metastases
Acronym: REVELATE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Blue Earth Diagnostics (Industry)
Collaborators: Precision For Medicine (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BED-FLC-312
Record Dates: First submitted 2020-05-27; First posted 2020-06-01 (Actual); Results first posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Brain Metastases
Keywords: Recurrent Brain Metastases; Diagnostic; Positron Emission Tomography (PET) Scan
MeSH Terms: conditions — Brain Neoplasms; Disease | interventions — fluciclovine F-18

STUDY DESIGN:
Intervention Model Description: Positron Emission Tomography (PET) Imaging study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Patients (Experimental): Single intravenous administration of 18F fluciclovine for PET Scan
  Interventions: Drug: 18F fluciclovine

INTERVENTIONS:
Drug: 18F fluciclovine — 18F fluciclovine injection, 185 MBq (5 mCi) ± 20%, delivered as an intravenous bolus
  Other Names: Axumin

SUMMARY:
An open-label, single dose, single arm, prospective, multicenter Phase 3 study to establish the diagnostic performance of 18F fluciclovine positron emission tomography (PET) in detecting recurrent brain metastases after radiation therapy

ELIGIBILITY:
Inclusion Criteria:

1. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1, or 2 if this is an acute deterioration
2. Previous history of solid tumor brain metastasis of any origin
3. Histopathological confirmation of the primary solid tumor or a metastatic site within 4 years
4. Previous radiation therapy of brain metastatic lesion(s)
5. A reference lesion considered by the site investigator to be equivocal for recurrent brain metastasis
6. Patient requires further confirmatory diagnostic procedures to confirm brain MRI findings and is planned for biopsy/neurosurgical intervention as standard of care (SoC) or clinical follow-up as SoC

Exclusion Criteria:

1. Patients with a history of active hematological malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2020-10-26 (Actual); Primary Completion 2023-06-05 (Actual); Study Completion 2023-06-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (19):
- United States (19):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - University of California, San Francisco, San Francisco, California
  - John Wayne Cancer Institute at Providence St. John's Health Center, Santa Monica, California
  - Yale School of Medicine, New Haven, Connecticut
  - Miami Cancer Institute at Baptist Health, Inc., Miami, Florida
  - Medical College of Georgia, Augusta University, Augusta, Georgia
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Johns Hopkins Hospital, Baltimore, Maryland
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Washington University School of Medicine-Center for Clinical Imaging Research, St Louis, Missouri
  - NYU Langone Health, New York, New York
  - University Hospital Cleveland, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Center for Quantitative Cancer Imaging at Huntsman Cancer Institute, Salt Lake City, Utah
  - West Virgina University Cancer Institute, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kotecha R, Aboian M, Nabavizadeh SA, Parent EE, Trifiletti DM, Chao ST. Letter regarding "Contribution of PET imaging to radiotherapy planning and monitoring in glioma patients-a report of the PET/RANO group": 18F-fluciclovine and target volume delineation. Neuro Oncol. 2021 Aug 2;23(8):1408-1409. doi: 10.1093/neuonc/noab097. No abstract available. PMID 34081125

RESULTS

PARTICIPANT FLOW:
Groups:
- Subjects Receiving Single IV Administration of 18F Fluciclovine for PET Scan: Subjects with a history of brain metastases previously treated with primary, adjuvant or repeat (salvage) radiation therapy, with a recent (within no more than 42 days before the study PET scan) SoC brain MRI found to be equivocal for recurrent brain metastasis, and who met all the inclusion criteria and none of the exclusion criteria, were consented and enrolled into the study. Specifically, subjects had to be planned for further confirmatory diagnostic procedures to confirm the brain MRI findings: either biopsy/neurosurgical intervention, or clinical follow-up, as SoC.
Period: Overall Study
Arm/Group | Subjects Receiving Single IV Administration of 18F Fluciclovine for PET Scan
Started | 151
Completed | 151
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Subjects Receiving Single IV Administration of 18F Fluciclovine for PET Scan
Number analyzed (Participants) | 151
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 81
  >=65 years | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.8 (11.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93
  Male | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18
  Not Hispanic or Latino | 131
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 134
  More than one race | 0
  Unknown or Not Reported | 4
Height (cm) [Mean (Standard Deviation); unit: cm] | 168.25 (10.002)
Weight (kg) [Mean (Standard Deviation); unit: kg] | 78.72 (19.665)
Body mass index (kg/m2) [Mean (Standard Deviation); unit: Kg/m2] | 27.66 (6.314)
ECOG [Count of Participants; unit: Participants] — ECOG performance status scale describes a patient's level of functioning:
  0=fully active, able to carry on as pre-disease without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light nature, e.g., light house work, office work
  2. Ambulatory/capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  3. Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours
  4. Completely disabled; cannot carry on any selfcare; totally confined to bed or chair
  Participants
    0 | 40
    1 | 96
    2 | 15
    3 | 0
    4 | 0

OUTCOME MEASURES:

1. Primary Outcome: Positive Percent Agreement (PPA) and Negative Percent Agreement (NPA) Subject Level
Description: Subject-level PPA and NPA (equivalent to sensitivity and specificity, respectively) of 18F-fluciclovinePET in detecting recurrent brain metastases.
Time Frame: MRI for anatomical correlation within 3 days of IMP and PET scan, followed by surgical intervention (if applicable) post-PET scan and follow up through 6 months after PET scan.
Measure: Number (95% Confidence Interval); unit: percentage
Groups:
- Reader 1 - Positive Percent Agreement (PPA); Reader 2 - Positive Percent Agreement (PPA); Reader 3 - Positive Percent Agreement (PPA): Only subjects with a positive standard of reference are included in the denominator for each reader.
- Reader 1 - Negative Percent Agreement (NPA); Reader 2 - Negative Percent Agreement (NPA); Reader 3 - Negative Percent Agreement (NPA): Only subjects with a negative standard of reference are included in the denominator for each reader.
Arm/Group | Reader 1 - Positive Percent Agreement (PPA) | Reader 2 - Positive Percent Agreement (PPA) | Reader 3 - Positive Percent Agreement (PPA) | Reader 1 - Negative Percent Agreement (NPA) | Reader 2 - Negative Percent Agreement (NPA) | Reader 3 - Negative Percent Agreement (NPA)
Number analyzed (Participants) | 42 | 41 | 41 | 109 | 110 | 110
percentage | 23.8 [12.1 to 39.5] | 34.1 [20.1 to 50.6] | 36.6 [22.1 to 53.1] | 82.6 [74.1 to 89.2] | 70.9 [61.5 to 79.2] | 70.9 [61.5 to 79.2]

2. Secondary Outcome: Subject Level Positive Predictive Value (PPV) and Negative Predictive Value (NPV)
Description: Subject-level PPV and NPV of 18F-fluciclovine PET for detecting recurrent brain metastases
Time Frame: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage
Groups:
- Reader 1 - Positive Predictive Value (PPV); Reader 2 - Positive Predictive Value (PPV); Reader 3 - Positive Predictive Value (PPV): Only subjects with a positive finding by BIE are included in the denominator for each reader.
- Reader 1 - Negative Predictive Value (NPV); Reader 2 - Negative Predictive Value (NPV); Reader 3 - Negative Predictive Value (NPV): Only subjects with a negative finding by BIE are included in the denominator for each reader.
Arm/Group | Reader 1 - Positive Predictive Value (PPV) | Reader 2 - Positive Predictive Value (PPV) | Reader 3 - Positive Predictive Value (PPV) | Reader 1 - Negative Predictive Value (NPV) | Reader 2 - Negative Predictive Value (NPV) | Reader 3 - Negative Predictive Value (NPV)
Number analyzed (Participants) | 29 | 46 | 47 | 122 | 105 | 104
percentage | 34.5 [17.9 to 54.3] | 30.4 [17.7 to 45.8] | 31.9 [19.1 to 47.1] | 73.8 [65.0 to 81.3] | 74.3 [64.8 to 82.5] | 75.0 [65.6 to 83.0]

3. Secondary Outcome: Lesion-level Positive Percent Agreement (PPA) and Negative Percent Agreement (NPA)
Description: To assess lesion-level PPA & NPA diagnostic performance of 18F-fluciclovine PET in detecting recurrent brain metastases.
Time Frame: as for outcome 1
Population: Each participant may have more than one lesion (one reference lesion, and/or other equivocal lesions and/or additional PET lesions if applicable). At the participant level, if the reference lesion is indeterminate, then the worst case is used to impute the indeterminate finding into positive or negative. However, at the lesion level, lesions with indeterminate findings are excluded i.e. only lesions with positive or negative finding are included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage
Units Other Than Participants: Lesions
Groups:
- Reader 1 - Positive Percent Agreement (PPA); Reader 2 - Positive Percent Agreement (PPA); Reader 3 - Positive Percent Agreement (PPA): Only Lesions with a positive standard of reference are included in the denominator for each reader.
- Reader 1 - Negative Percent Agreement (NPA); Reader 2 - Negative Percent Agreement (NPA); Reader 3 - Negative Percent Agreement (NPA): Only Lesions with a negative standard of reference are included in the denominator for each reader.
Arm/Group | Reader 1 - Positive Percent Agreement (PPA) | Reader 2 - Positive Percent Agreement (PPA) | Reader 3 - Positive Percent Agreement (PPA) | Reader 1 - Negative Percent Agreement (NPA) | Reader 2 - Negative Percent Agreement (NPA) | Reader 3 - Negative Percent Agreement (NPA)
Number analyzed (Participants) | 42 | 41 | 41 | 109 | 110 | 110
Number analyzed (Lesions) | 49 | 49 | 49 | 138 | 138 | 138
percentage | 18.4 [7.3 to 29.4] | 28.6 [15.8 to 41.4] | 30.6 [17.7 to 43.5] | 84.1 [77.4 to 90.7] | 74.6 [66.6 to 82.7] | 73.2 [65.0 to 81.4]

4. Secondary Outcome: Lesion-level Positive Predictive Value (PPV) and Negative Predictive Value (NPV)
Description: To assess lesion-level PPV & NPV diagnostic performance of 18F-fluciclovine PET in detecting recurrent brain metastases.
Time Frame: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage
Units Other Than Participants: Lesions
Groups:
- Reader 1 - Positive Predictive Value (PPV); Reader 2 - Positive Predictive Value (PPV); Reader 3 - Positive Predictive Value (PPV): Only Lesions with a positive finding by BIE are included in the denominator for reach reader
- Reader 1 - Negative Predictive Value (NPV); Reader 2 - Negative Predictive Value (NPV); Reader 3 - Negative Predictive Value (NPV): Only Lesions with a negative finding by BIE are included in the denominator for reach reader
Arm/Group | Reader 1 - Positive Predictive Value (PPV) | Reader 2 - Positive Predictive Value (PPV) | Reader 3 - Positive Predictive Value (PPV) | Reader 1 - Negative Predictive Value (NPV) | Reader 2 - Negative Predictive Value (NPV) | Reader 3 - Negative Predictive Value (NPV)
Number analyzed (Participants) | 29 | 46 | 47 | 122 | 105 | 104
Number analyzed (Lesions) | 31 | 49 | 52 | 156 | 138 | 135
percentage | 29.0 [12.1 to 45.9] | 28.6 [15.2 to 42.0] | 28.8 [15.3 to 42.4] | 74.4 [65.5 to 83.2] | 74.6 [65.4 to 83.9] | 74.8 [65.8 to 83.8]

5. Secondary Outcome: Subject-level Positive Percent Agreement (PPA) & Negative Percent Agreement (NPA) Diagnostic Performance of Fluciclovine (18F) PET in Detecting Recurrent Brain Metastases in Different Clinical Settings - Tumor Type
Description: Sub-group analyses of subject-level PPA & NPA of fluciclovine (18F) PET, according to primary tumor type.
Time Frame: as for outcome 1
Population: All subjects with a positive or negative Standard of Reference (SoR), with outcome measures categorized by tumor type.
Measure: Number (95% Confidence Interval); unit: percentage
Groups:
- Reader 1 - Positive Percent Agreement (NPA); Reader 2 - Positive Percent Agreement (NPA); Reader 3 - Positive Percent Agreement (NPA): Only subjects with a positive standard of reference are included in the denominator for each reader.
Arm/Group | Reader 1 - Positive Percent Agreement (NPA) | Reader 2 - Positive Percent Agreement (NPA) | Reader 3 - Positive Percent Agreement (NPA) | Reader 1 - Negative Percent Agreement (NPA) | Reader 2 - Negative Percent Agreement (NPA) | Reader 3 - Negative Percent Agreement (NPA)
Number analyzed (Participants) | 42 | 41 | 41 | 109 | 110 | 110
percentage
  Melanoma: number analyzed (Participants) | 2 | 2 | 2 | 18 | 18 | 18
  Melanoma | 50.0 [1.3 to 98.7] | 50.0 [1.3 to 98.7] | 0.0 [0.0 to 84.2] | 83.3 [58.6 to 96.4] | 72.2 [46.5 to 90.3] | 66.7 [41.0 to 86.7]
  Breast: number analyzed (Participants) | 10 | 10 | 10 | 23 | 23 | 23
  Breast | 10.0 [0.3 to 44.5] | 30.0 [6.7 to 65.3] | 40.0 [12.2 to 73.8] | 78.3 [56.3 to 92.5] | 65.2 [42.7 to 83.6] | 73.9 [51.6 to 89.8]
  Lung Cancer: number analyzed (Participants) | 24 | 23 | 23 | 48 | 49 | 49
  Lung Cancer | 29.2 [12.6 to 51.1] | 39.1 [19.7 to 61.5] | 43.5 [23.2 to 65.5] | 85.4 [72.2 to 93.9] | 69.4 [54.6 to 81.8] | 67.3 [52.5 to 80.1]
  Non Lung/Breast/Melanoma: number analyzed (Participants) | 6 | 6 | 6 | 20 | 20 | 20
  Non Lung/Breast/Melanoma | 16.7 [0.4 to 64.1] | 16.7 [0.4 to 64.1] | 16.7 [0.4 to 64.1] | 80.0 [56.3 to 94.3] | 80.0 [56.3 to 94.3] | 80.0 [56.3 to 94.3]

6. Secondary Outcome: Subject-level Positive Predictive Value (PPV) & Negative Predictive Value (NPV) Diagnostic Performance of Fluciclovine (18F) PET in Detecting Recurrent Brain Metastases in Different Clinical Settings - Tumor Type
Description: Sub-group analyses of subject-level PPV & NPV of fluciclovine (18F) PET, according to primary tumor type.
Time Frame: as for outcome 1
Population: All subjects with a positive or negative finding by BIE, with outcome measures categorized by tumor type.
Measure: Number (95% Confidence Interval); unit: percentage
Groups:
- Reader 1 - Positive Predictive Value (PPV); Reader 2 - Positive Predictive Value (PPV); Reader 3 - Positive Predictive Value (PPV): Only subjects with a positive finding by BIE are included in the denominator for reach reader
- Reader 1 - Negative Predictive Value (NPV); Reader 2 - Negative Predictive Value (NPV); Reader 3 - Negative Predictive Value (NPV): Only subjects with a negative finding by BIE are included in the denominator for reach reader
Arm/Group | Reader 1 - Positive Predictive Value (PPV) | Reader 2 - Positive Predictive Value (PPV) | Reader 3 - Positive Predictive Value (PPV) | Reader 1 - Negative Predictive Value (NPV) | Reader 2 - Negative Predictive Value (NPV) | Reader 3 - Negative Predictive Value (NPV)
Number analyzed (Participants) | 29 | 46 | 47 | 122 | 105 | 104
percentage
  Melanoma: number analyzed (Participants) | 4 | 6 | 6 | 16 | 14 | 14
  Melanoma | 25.0 [0.6 to 80.6] | 16.7 [0.4 to 64.1] | 0.0 [0.0 to 45.9] | 93.8 [69.8 to 99.8] | 92.9 [66.1 to 99.8] | 85.7 [57.2 to 98.2]
  Breast: number analyzed (Participants) | 6 | 11 | 10 | 27 | 22 | 23
  Breast | 16.7 [0.4 to 64.1] | 27.3 [6.0 to 61.0] | 40.0 [12.2 to 73.8] | 66.7 [46.0 to 83.5] | 68.2 [45.1 to 86.1] | 73.9 [51.6 to 89.8]
  Lung Cancer: number analyzed (Participants) | 14 | 24 | 26 | 58 | 48 | 46
  Lung Cancer | 50.0 [23.0 to 77.0] | 37.5 [18.8 to 59.4] | 38.5 [20.2 to 59.4] | 70.7 [57.3 to 81.9] | 70.8 [55.9 to 83.1] | 71.7 [56.5 to 84.0]
  Non Lung/Breast/Melanoma: number analyzed (Participants) | 5 | 5 | 5 | 21 | 21 | 21
  Non Lung/Breast/Melanoma | 20.0 [0.5 to 71.6] | 20.0 [0.5 to 71.6] | 20.0 [0.5 to 71.6] | 76.2 [52.8 to 91.8] | 76.2 [52.8 to 91.8] | 76.2 [52.8 to 91.8]

7. Secondary Outcome: Subject-level Positive Percent Agreement (NPA) & Negative Percent Agreement (NPA) Diagnostic Performance of Fluciclovine (18F) PET in Detecting Recurrent Brain Metastases in Different Clinical Settings - Concurrent Immunotherapy
Description: Sub-group analyses of subject-level PPA & NPA of fluciclovine (18F) PET, according to concurrent immunotherapy.
Time Frame: as for outcome 1
Population: All subjects with a positive or negative Standard of Reference (SoR), with outcome measures categorized by concurrent Immunotherapy.
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Reader 1 - Positive Percent Agreement (NPA) | Reader 2 - Positive Percent Agreement (NPA) | Reader 3 - Positive Percent Agreement (NPA) | Reader 1 - Negative Percent Agreement (NPA) | Reader 2 - Negative Percent Agreement (NPA) | Reader 3 - Negative Percent Agreement (NPA)
Number analyzed (Participants) | 42 | 41 | 41 | 109 | 110 | 110
percentage
  Received Concurrent Immunotherapy: number analyzed (Participants) | 6 | 6 | 6 | 30 | 30 | 30
  Received Concurrent Immunotherapy | 0.0 [0.0 to 45.9] | 16.7 [0.4 to 64.1] | 16.7 [0.4 to 64.1] | 100.0 [88.4 to 100.0] | 86.7 [69.3 to 96.2] | 90.0 [73.5 to 97.9]
  Did Not Receive Concurrent Immunotherapy: number analyzed (Participants) | 36 | 35 | 35 | 79 | 80 | 80
  Did Not Receive Concurrent Immunotherapy | 27.8 [14.2 to 45.2] | 37.1 [21.5 to 55.1] | 40.0 [23.9 to 57.9] | 75.9 [65.0 to 84.9] | 65.0 [53.5 to 75.3] | 63.8 [52.2 to 74.2]

8. Secondary Outcome: Subject-level Positive Predictive Value (PPV) & Negative Predictive Value (NPV) Diagnostic Performance of Fluciclovine (18F) PET in Detecting Recurrent Brain Metastases in Different Clinical Settings - Concurrent Immunotherapy
Description: Sub-group analyses of subject-level PPV & NPV of fluciclovine (18F) PET, according to Concurrent Immunotherapy.
Time Frame: as for outcome 1
Population: All subjects with a positive or negative finding by BIE, with outcome measures categorized by concurrent Immunotherapy.
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Reader 1 - Positive Predictive Value (PPV) | Reader 2 - Positive Predictive Value (PPV) | Reader 3 - Positive Predictive Value (PPV) | Reader 1 - Negative Predictive Value (NPV) | Reader 2 - Negative Predictive Value (NPV) | Reader 3 - Negative Predictive Value (NPV)
Number analyzed (Participants) | 29 | 46 | 47 | 122 | 105 | 104
percentage
  Received Concurrent Immunotherapy: number analyzed (Participants) | 0 | 5 | 4 | 36 | 31 | 32
  Received Concurrent Immunotherapy |  | 20.0 [0.5 to 71.6] | 25.0 [0.6 to 80.6] | 83.3 [67.2 to 93.6] | 83.9 [66.3 to 94.6] | 84.4 [67.2 to 94.7]
  Did Not Receive Concurrent Immunotherapy: number analyzed (Participants) | 29 | 41 | 43 | 86 | 74 | 72
  Did Not Receive Concurrent Immunotherapy | 34.5 [17.9 to 54.3] | 31.7 [18.1 to 48.1] | 32.6 [19.1 to 48.5] | 69.8 [58.9 to 79.2] | 70.3 [58.5 to 80.3] | 70.8 [58.9 to 81.0]

9. Secondary Outcome: Clinical Usefulness
Description: Number of days taken by the site to establish presence/absence of metastasis by clinical follow-up.
Time Frame: Follow up through 6 months after PET scan.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Subjects Receiving Single IV Administration of 18F Fluciclovine for PET Scan
Number analyzed (Participants) | 151
Days | 112 [77.0 to 142.0]

10. Secondary Outcome: Clinical Usefulness
Description: Proportion of subjects with additional metastases identified on fluciclovine (18F) PET in addition to SoC brain MRI
Time Frame: Follow up through 6 months after PET scan.
Population: Subjects with Additional Metastases Identified on Fluciclovine (18F) PET vs SoC MRI
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Subjects Receiving Single IV Administration of 18F Fluciclovine for PET Scan
Number analyzed (Participants) | 151
percentage | 1.3 [0.2 to 4.7]

11. Secondary Outcome: Clinical Usefulness
Description: Proportion of subjects whose prospective diagnostic management plan changed following fluciclovine (18F) PET.
Time Frame: Follow up through 6 months after PET scan.
Population: Subjects with Changes to Diagnostic Plan on Reference Lesion Following Fluciclovine (18F) PET
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Subjects Receiving Single IV Administration of 18F Fluciclovine for PET Scan
Number analyzed (Participants) | 151
percentage | 26.5 [19.7 to 34.3]

12. Secondary Outcome: Inter-reader Reproducibility
Description: Pairwise comparisons of the central reads for the 3 readers (i.e. Reader 1 vs Reader 2, Reader 1 vs Reader 3, and Reader 2 vs Reader 3) at the subject-level. The percentage of results in agreement (i.e. Positive [1st reader] / Positive [2nd reader], Negative/Negative) is presented.
Time Frame: PET Scan Day 1
Measure: Number; unit: percentage
Arm/Group | Subjects Receiving Single IV Administration of 18F Fluciclovine for PET Scan
Number analyzed (Participants) | 151
percentage
  Reader 1 vs Reader 2 | 86.1
  Reader 1 vs Reader 3 | 84.1
  Reader 2 vs Reader 3 | 91.4

13. Secondary Outcome: Intra-reader Reproducibility
Description: Pairwise comparisons of the initial read vs re-read of a subset of PET scans for each reader at the subject-level. The percentage of results in agreement (i.e. Positive [initial read] / Positive [re-read], Negative/Negative) is presented.
Time Frame: PET Scan Day 1
Measure: Number; unit: percentage
Arm/Group | Subjects Receiving Single IV Administration of 18F Fluciclovine for PET Scan
Number analyzed (Participants) | 31
percentage
  Reader 1 initial read vs re-read | 93.5
  Reader 2 initial read vs re-read | 93.5
  Reader 3 initial read vs re-read | 100.0

14. Secondary Outcome: Assess the Safety of Fluciclovine (18F) Injection in the Subject Population, Blood Pressure
Description: Treatment-emergent adverse events (TEAEs) following 18F-fluciclovine injection in the subject population.
Time Frame: The vital signs collected between 5 to 60 minutes before and after the PET scan.
Population: Collected and Reported
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Subjects Receiving Single IV Administration of 18F Fluciclovine for PET Scan
Number analyzed (Participants) | 151
mmHg
  Systolic Blood Pressure: Pre-IMP Injection: number analyzed (Participants) | 145
  Systolic Blood Pressure: Pre-IMP Injection | 128.7 (17.25)
  Systolic Blood Pressure: Post PET Scan: number analyzed (Participants) | 145
  Systolic Blood Pressure: Post PET Scan | 132.4 (15.25)
  Systolic Blood Pressure: Change from Pre to Post: number analyzed (Participants) | 144
  Systolic Blood Pressure: Change from Pre to Post | 3.5 (12.81)
  Diastolic Blood Pressure: Pre-IMP Injection: number analyzed (Participants) | 145
  Diastolic Blood Pressure: Pre-IMP Injection | 75.4 (10.69)
  Diastolic Blood Pressure: Post PET Scan: number analyzed (Participants) | 145
  Diastolic Blood Pressure: Post PET Scan | 77.0 (10.86)
  Diastolic Blood Pressure: Change from Pre to Post: number analyzed (Participants) | 144
  Diastolic Blood Pressure: Change from Pre to Post | 1.5 (7.45)

15. Secondary Outcome: Assess the Safety of Fluciclovine (18F) Injection in the Subject Population, Heart Rate
Description: Treatment-emergent adverse events (TEAEs) following 18F-fluciclovine injection in the subject population.
Time Frame: The vital signs collected between 5 to 60 minutes before and after the PET scan.
Population: Collected and Reported
Measure: Mean (Standard Deviation); unit: beat/min
Arm/Group | Subjects Receiving Single IV Administration of 18F Fluciclovine for PET Scan
Number analyzed (Participants) | 151
beat/min
  Heart Rate: Pre-IMP Injection: number analyzed (Participants) | 144
  Heart Rate: Pre-IMP Injection | 76.2 (13.53)
  Heart Rate: Post PET Scan: number analyzed (Participants) | 144
  Heart Rate: Post PET Scan | 74.5 (12.93)
  Heart Rate: Change from Pre to Post: number analyzed (Participants) | 144
  Heart Rate: Change from Pre to Post | -1.7 (8.43)

16. Secondary Outcome: Assess the Safety of Fluciclovine (18F) Injection in the Subject Population, Respiratory Rate
Description: Treatment-emergent adverse events (TEAEs) following 18F-fluciclovine injection in the subject population.
Time Frame: The vital signs collected between 5 to 60 minutes before and after the PET scan.
Population: Collected and Reported
Measure: Mean (Standard Deviation); unit: breaths/min
Arm/Group | Subjects Receiving Single IV Administration of 18F Fluciclovine for PET Scan
Number analyzed (Participants) | 151
breaths/min
  Respiratory Rate: Pre-IMP Injection: number analyzed (Participants) | 143
  Respiratory Rate: Pre-IMP Injection | 16.7 (2.76)
  Respiratory Rate: Post PET Scan: number analyzed (Participants) | 141
  Respiratory Rate: Post PET Scan | 16.5 (2.72)
  Respiratory Rate: Change from Pre to Post: number analyzed (Participants) | 141
  Respiratory Rate: Change from Pre to Post | -0.2 (1.85)

17. Secondary Outcome: Assess the Safety of Fluciclovine (18F) Injection in the Subject Population, Body Temperature
Description: Treatment-emergent adverse events (TEAEs) following 18F-fluciclovine injection in the subject population.
Time Frame: The vital signs collected between 5 to 60 minutes before and after the PET scan.
Population: Collected and Reported
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | Subjects Receiving Single IV Administration of 18F Fluciclovine for PET Scan
Number analyzed (Participants) | 151
degrees Celsius
  Body Temperature: Pre-IMP Injection: number analyzed (Participants) | 141
  Body Temperature: Pre-IMP Injection | 36.53 (0.419)
  Body Temperature: Post PET Scan: number analyzed (Participants) | 142
  Body Temperature: Post PET Scan | 36.53 (0.455)
  Body Temperature: Change from Pre to Post: number analyzed (Participants) | 142
  Body Temperature: Change from Pre to Post | -0.00 (0.29)

ADVERSE EVENTS:
Time Frame: Treatment emerging AEs were captured within 48 hours.
Arm/Group | Subjects Receiving Single IV Administration of 18F Fluciclovine for PET Scan
All-Cause Mortality (participants affected / at risk) | 0/151
Serious Adverse Events (participants affected / at risk) | 2/151
Other Adverse Events (participants affected / at risk) | 15/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects Receiving Single IV Administration of 18F Fluciclovine for PET Scan (N=151)
Seizure (Nervous system disorders) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects Receiving Single IV Administration of 18F Fluciclovine for PET Scan (N=151)
Fatigue (General disorders) | 4 (4)
Infusion site bruising (General disorders) | 1 (1)
Injection site reaction (General disorders) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Hordeolum (Infections and infestations) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-03-17): https://cdn.clinicaltrials.gov/large-docs/33/NCT04410133/Prot_002.pdf
  • Statistical Analysis Plan (2021-07-13): https://cdn.clinicaltrials.gov/large-docs/33/NCT04410133/SAP_003.pdf